CLINICAL TRIAL: NCT04254965
Title: Music Therapy Intervention and Bio-psychological Effects Evaluation Among Chronic Psychiatric Inpatients in Rehabilitation Wards of a Community Teaching Hospital
Brief Title: Music Therapy and Bio-psychological Effect Among Chronic Psychiatric Inpatients of a Community Teaching Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Tsing Hua University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 201908035RINC
Record Dates: First submitted 2020-01-05; First posted 2020-02-05 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Chronic Psychosis
Keywords: music therapy; chronic psychosis; negative symptoms; occupational therapy; biosignal analysis
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group 1 (Experimental): Participants of integrated music therapy (integration of active and passive music therapy) includes instrument playing, singing, lyrics modification/music organized play, listening to music and discussing each treatment process. The four stages of activities are warm-up, main activities, secondary activities, and the ending section.
  Interventions: Other: Music therapy; Device: Biosignal analysis
- Group 2 (Active Comparator): Participants of the music listening group will receive background music listening, music selection based on the musical preference and background of subjects, for relax or boost the spirit of the subjects.
  Interventions: Other: Music therapy; Device: Biosignal analysis
- Group 3 (Sham Comparator): Participants in the control group receive their regular occupational therapy during the experimental period.
  Interventions: Device: Biosignal analysis

INTERVENTIONS:
Other: Music therapy — Treatment including instrument playing, singing, lyrics modification/music organized play, listening to music and discussing each treatment process.
  Arms: Group 1; Group 2
Device: Biosignal analysis — Measurement of facial expression emotion recognition, electrodermal activity, heart rate variability, sleep pattern, blood pressure, and electromyogram.
  Other Names: iMotions; GSR-Shimmer Module; Dailycare; Fitbit; DELYSYS TrignoTM Flex

SUMMARY:
Negative symptoms are an important factor in preventing patients from returning to the community, we aim to assess the effect of music therapy on negative symptoms through this study. Participants of integrated music therapy will receive instrument playing, singing, lyrics modification/music organized play, listening to music and discussing each treatment process. Other participants will receive passive music listening or regular occupational therapy during the experimental period. Psychiatric symptoms, quality of life, social and interactive skills, and the differences in the physiological signals produced by skin, muscles, and heart will be measured before, after, and two months after the music therapy.

DETAILED DESCRIPTION:
Music therapy is gradually being used in the field of psychiatry, such as depression, anxiety, and development disorders in children. However, music therapy still lacks systematic research on chronic mental illness. Since negative symptoms are an important factor in preventing patients from returning to the community, we aim to assess the effect of music therapy on negative symptoms through this study. Additionally, Taiwan as many Asian countries have not yet established a certification system for music therapy. This study cooperates with licensed therapists abroad in the hope of promoting the systematic development of local music therapy in the future.

Participants of integrated music therapy (Group 1, integration of active and passive music therapy) includes instrument playing, singing, lyrics modification/music organized play, listening to music and discussing each treatment process. The four stages of activities are warm-up, main activities, secondary activities, and the ending section. The participants of the music listening group (Group 2, background music listening), music selection based on the musical preference and background of subjects, for relax or boost the spirit of the subjects. Participants in the control group (Group 3) receive their regular occupational therapy during the experimental period. We plan to recruit 100 people in the wards: 40/20/40 (Group 1/2/3) under random assignment.

To evaluate the effects of three groups, we measure their psychiatric symptoms, quality of life, social and interactive skills, and the differences in the physiological signals produced by skin, muscles, and heart assisted by a medical engineering scholar before, after, and two months after the music therapy.

ELIGIBILITY:
Inclusion criteria

* Chronic patient in rehabilitation ward without compulsory hospitalization.
* Patients with mental, behavioral and neurodevelopmental disorders, including schizophrenia, schizotypal personality disorders, delusional disorders, affective disorders, and organic mental disorders.

Exclusion criteria

* Patients with hearing impairments.
* Patients with no capacity to make juridical acts.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change of negative symptoms of inpatients with psychotic disorders | Before and immediately after finishing the music therapy
  Using the Scale for the Assessment of Negative Symptoms (in Traditional Chinese)
Change of negative symptoms of inpatients with psychotic disorders | Before and 2 months after finishing the music therapy
  Using the Scale for the Assessment of Negative Symptoms (in Traditional Chinese)
Change of quality of life | Before and immediately after finishing the music therapy
  Using the World Health Organization Quality of Life-BREF questionnaire (it is a compress name, Traditional Chinese version). The WHOQOL-BREF was derived from data collected using the WHOQOL-100. It produces scores for four domains related to quality of life: physical health, psychological, social relationships and environment. It also includes one facet on overall quality of life and general health. Potential scores for all domain scores range from 4(worse) to 20(better).
Change of quality of life | Before and 2 months after finishing the music therapy
  Using the World Health Organization Quality of Life-BREF questionnaire (it is a compress name, Traditional Chinese version). The WHOQOL-BREF was derived from data collected using the WHOQOL-100. It produces scores for four domains related to quality of life: physical health, psychological, social relationships and environment. It also includes one facet on overall quality of life and general health. Potential scores for all domain scores range from 4(worse) to 20(better).
Change of social and interactive skills | Before and immediately after finishing the music therapy
  Using the Assessment of Communication and Interaction Skills scale (in Traditional Chinese)
Change of social and interactive skills | Before and 2 months after finishing the music therapy
  Using the Assessment of Communication and Interaction Skills scale (in Traditional Chinese)

SECONDARY OUTCOMES:
Change of facial expression by action landmarks | Two months
  To evaluate emotion (e.g. anger, fear, disgust, contempt, sadness, and surprise) via facial motion by iMotions device
Heart Rate Variability in Psychiatric Disorders analysis | Two months
  Measure Heartbeat variability after intervention activities by "Dailycare" CheckMyHeart
Total sleeping time | Two months
  Recorded by Fitbit health watch
Sleep schedule | Two months
  Recorded by Fitbit health watch, meaning the hours patients are asleep
Sleep pattern | Two months
  Recorded by Fitbit health watch, meaning the distribution of sleep stages (light sleep, deep sleep and rapid eye movement sleep).
Motion analysis | Two months
  Analysis of the electromyography (EMG) of cases recorded by DELYSYS, EMG potentials range between less than 50 μV and up to 30 mV.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Che Chen, MDMPH, Principal Investigator — National Taiwan University Hospital Chu-Tung Branch
Locations (1):
- National Taiwan University Hospital, Hsinchu, Hsinchu County, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gold C, Rolvsjord R, Aaro LE, Aarre T, Tjemsland L, Stige B. Resource-oriented music therapy for psychiatric patients with low therapy motivation: protocol for a randomised controlled trial [NCT00137189]. BMC Psychiatry. 2005 Oct 31;5:39. doi: 10.1186/1471-244X-5-39. PMID 16259626
- [Background] Buccheri R, Trygstad L, Dowling G, Hopkins R, White K, Griffin JJ, Henderson S, Suciu L, Hippe S, Kaas MJ, Covert C, Hebert P. Long-term effects of teaching behavioral strategies for managing persistent auditory hallucinations in schizophrenia. J Psychosoc Nurs Ment Health Serv. 2004 Jan;42(1):18-27. doi: 10.3928/02793695-20040101-09. PMID 14768276
- [Background] Acil AA, Dogan S, Dogan O. The effects of physical exercises to mental state and quality of life in patients with schizophrenia. J Psychiatr Ment Health Nurs. 2008 Dec;15(10):808-15. doi: 10.1111/j.1365-2850.2008.01317.x. PMID 19012672
- [Background] Cook JD. Music as an intervention in the oncology setting. Cancer Nurs. 1986 Feb;9(1):23-8. No abstract available. PMID 3518914
- [Background] Wiersma D, Jenner JA, Nienhuis FJ, van de Willige G. Hallucination focused integrative treatment improves quality of life in schizophrenia patients. Acta Psychiatr Scand. 2004 Mar;109(3):194-201. doi: 10.1046/j.0001-690x.2003.00237.x. PMID 14984391
- [Background] Morgan KA, Harris AW, Luscombe G, Tran Y, Herkes G, Bartrop RW. The effect of music on brain wave functioning during an acute psychotic episode: a pilot study. Psychiatry Res. 2010 Jul 30;178(2):446-8. doi: 10.1016/j.psychres.2010.04.020. Epub 2010 May 14. PMID 20471105
- [Background] Silverman MJ. Psychiatric patients' perception of music therapy and other psychoeducational programming. J Music Ther. 2006 Summer;43(2):111-22. doi: 10.1093/jmt/43.2.111. PMID 16897904
- [Background] Peng SM, Koo M, Kuo JC. Effect of group music activity as an adjunctive therapy on psychotic symptoms in patients with acute schizophrenia. Arch Psychiatr Nurs. 2010 Dec;24(6):429-34. doi: 10.1016/j.apnu.2010.04.001. Epub 2010 May 21. PMID 21111297
- [Background] Ulrich G, Houtmans T, Gold C. The additional therapeutic effect of group music therapy for schizophrenic patients: a randomized study. Acta Psychiatr Scand. 2007 Nov;116(5):362-70. doi: 10.1111/j.1600-0447.2007.01073.x. PMID 17919155
- [Background] Hayashi N, Tanabe Y, Nakagawa S, Noguchi M, Iwata C, Koubuchi Y, Watanabe M, Okui M, Takagi K, Sugita K, Horiuchi K, Sasaki A, Koike I. Effects of group musical therapy on inpatients with chronic psychoses: a controlled study. Psychiatry Clin Neurosci. 2002 Apr;56(2):187-93. doi: 10.1046/j.1440-1819.2002.00953.x. PMID 11952923
- [Background] Chou MH, Lin MF. Exploring the listening experiences during guided imagery and music therapy of outpatients with depression. J Nurs Res. 2006 Jun;14(2):93-102. doi: 10.1097/01.jnr.0000387567.41941.14. PMID 16741859
- [Background] Talwar N, Crawford MJ, Maratos A, Nur U, McDermott O, Procter S. Music therapy for in-patients with schizophrenia: exploratory randomised controlled trial. Br J Psychiatry. 2006 Nov;189:405-9. doi: 10.1192/bjp.bp.105.015073. PMID 17077429
- [Background] Hars M, Herrmann FR, Gold G, Rizzoli R, Trombetti A. Effect of music-based multitask training on cognition and mood in older adults. Age Ageing. 2014 Mar;43(2):196-200. doi: 10.1093/ageing/aft163. Epub 2013 Nov 7. PMID 24212920
- [Background] Tseng PT, Chen YW, Lin PY, Tu KY, Wang HY, Cheng YS, Chang YC, Chang CH, Chung W, Wu CK. Significant treatment effect of adjunct music therapy to standard treatment on the positive, negative, and mood symptoms of schizophrenic patients: a meta-analysis. BMC Psychiatry. 2016 Jan 26;16:16. doi: 10.1186/s12888-016-0718-8. Erratum In: BMC Psychiatry. 2016 May 17;16:150. doi: 10.1186/s12888-016-0846-1. PMID 26812906